CLINICAL TRIAL: NCT02036593
Title: Community Approaches to Cardiovascular Health: Pathways to Heart Health (CATCH-PATH)
Brief Title: Community Approaches to Cardiovascular Health: Pathways to Heart Health
Acronym: CATCH-PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Amy J. Schulz, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CATCH-PATH; 2R24MD001619-04 (NIH)
Record Dates: First submitted 2013-12-17; First posted 2014-01-15 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Cardiovascular Risk Factors
Keywords: Cardiovascular Risk Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Walk Your Heart to Health intervention (Experimental): Participants were randomized into one of two groups: intervention and lagged intervention. The intervention group completed the 8 week Walk Your Heart to Health intervention, followed by a second wave of data collection for both initial and lagged intevention groups. The lagged intervention group then completed the 8 week Walk Your Heart to Health intervention. Both groups continued walking for another 24 weeks.
  Walking group sessions conducted 3 times per week for 32 weeks.
  Interventions: Behavioral: Walk Your Heart to Health
- Walk Your Heart to Health lagged (Other): Participants were randomized into one of two groups: intervention and lagged intervention. The intervention group completed the 8 week Walk Your Heart to Health intervention, followed by a second wave of data collection for both initial and lagged intevention groups. The lagged intervention group then completed the 8 week Walk Your Heart to Health intervention. Both groups continued walking for another 24 weeks.
  Walking group sessions conducted 3 times per week for 32 weeks.
  Interventions: Behavioral: Walk Your Heart to Health

INTERVENTIONS:
Behavioral: Walk Your Heart to Health — Walking group sessions conducted 3 times per week for 32 weeks.

SUMMARY:
The Specific Aims for CATCH: PATH are:

Specific Aim 1: To promote cardiovascular health through implementation and evaluation of a multilevel CBPR intervention (i.e., individual, family, organizational levels) to increase opportunities for active living, specifically walking groups, in three communities in Detroit.

Specific Aim 2: To promote cardiovascular health through implementation and evaluation of a multilevel CBPR intervention (i.e., organization, community, policy levels) to promote leadership development, community action, and policy level change to enhance neighborhood environments that support and sustain active living.

Specific Aim 3: To maintain and evaluate the HEP CBPR partnership engaging members of the partnership in providing scientific and community oversight for all aspects of the CATCH: PATH project.

Specific Aim 4: To disseminate preliminary results and develop a comprehensive Dissemination Plan to share research findings through community and peer reviewed outlets to assure translation of results from this multilevel CBPR intervention into programmatic and policy efforts to improve heart health in eastside, northwest and southwest Detroit.

DETAILED DESCRIPTION:
The Specific Aims for CATCH: PATH are:

Specific Aim 1: To promote cardiovascular health through implementation and evaluation of a multilevel CBPR intervention (i.e., individual, family, organizational levels) to increase opportunities for active living, specifically walking groups, in three communities in Detroit.

Specific Aim 2: To promote cardiovascular health through implementation and evaluation of a multilevel CBPR intervention (i.e., organization, community, policy levels) to promote leadership development, community action, and policy level change to enhance neighborhood environments that support and sustain active living.

Specific Aim 3: To maintain and evaluate the HEP CBPR partnership engaging members of the partnership in providing scientific and community oversight for all aspects of the CATCH: PATH project.

Specific Aim 4: To disseminate preliminary results and develop a comprehensive Dissemination Plan to share research findings through community and peer reviewed outlets to assure translation of results from this multilevel CBPR intervention into programmatic and policy efforts to improve heart health in eastside, northwest and southwest Detroit.

Research Questions and Hypotheses

In Aim 1, we intend to assess the short term (8 week) and longer term (10 month) effectiveness of a multilevel CBPR intervention (i.e., individual, family, organizational levels) designed to improve heart health through enhanced opportunities for active living, specifically walking groups, in three communities in Detroit. Hypotheses to be tested are:

Participation in an 8-week intensive walking group intervention will reduce risk factors and increase protective factors associated with CVD among African American, Latino and white residents of low to moderate income neighborhoods in Detroit.

H1.1: Physical activity will increase (physical inactivity will be reduced). H1.2: Psychosocial factors positively associated with physical activity (e.g., confidence in ability to be physically active most days of the week) will increase.

H1.3: Anthropometric indicators of CVD risk (e.g., BMI, waist circumference) will not change significantly.

H1.4: Biological indicators of CVD risk (e.g., lipid levels) will not change significantly.

Participation in a less intensive, maintenance walking group intervention over a 10 month period following the initial intensive walking groups will sustain changes in physical activity, further improvements in psychosocial factors associated with reduced risk, and reductions in biological and anthropomorphic risk factors and improvements in protective factors among participants.

H2.1: Increases in physical activity from baseline will be sustained during the maintenance period (physical inactivity will be reduced from baseline).

H2.2: Increases in psychosocial factors positively associated with physical activity (e.g., confidence in ability to be physically active most days of the week) will be enhanced (improved at 12 months over baseline and over the immediate post-intervention follow up).

H2.3: Anthropometric indicators of CVD risk (e.g., BMI, waist circumference) will be reduced at 12 months compared to baseline.

H2.4: Biological indicators of CVD risk (e.g., LDL levels) will be reduced and protective indicators (e.g., HDL) increased at 12 months compared to baseline.

In Aim 2, we will assess the feasibility of promoting heart health by providing support for leadership development, organizational change, community action and policy change to enhance neighborhood environments that support and sustain active living. Research questions will examine: the extent to which provision of technical assistance and facilitator training to community organizations can support the development and maintenance of walking groups and the extent to which a mini-grant program contributes to modifications of the built and social environment to support active living. These exploratory research questions, essential to the dissemination and sustainability of community-based interventions addressing disparities in CVD, will not be tested as formal hypotheses. Rather, we will focus on documenting change, and identifying challenges, facilitating factors, and lessons learned to inform subsequent more formal hypotheses-testing.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years old and over
* Residents of Detroit, MI

Exclusion Criteria:

* Individual has a legal guardian
* Individual is pregnant and delivery is expected within the next 5 months
* Individual answers yes to any of the following questions on a screening questionnaire and DOES NOT provide a medical clearance from his/her physician:

  1. Has your doctor ever said that you have a heart condition and that you should only do physical activity recommended by a doctor?
  2. Do you feel pain in your chest when you do physical activity?
  3. In the past month, have you had chest pain when you were not doing physical activity?
  4. Do you lose your balance because of dizziness or do you ever lose consciousness?
  5. Do you have a bone or joint problem that could be made worse by a change in physical activity?
  6. Do you have type I diabetes, sometimes called juvenile onset diabetes?
  7. Has your doctor advised you NOT to participate in exercise because of any of the above reasons?
  8. Are you aware, through your own experience or doctors advice, of any other physical reason which would prevent you from exercising without medical supervision or specific instructions from a doctor?

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 695 (Actual)
Dates: Start 2008-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pedometer steps | Pedometer data will be uploaded for each participant at each session, at least weekly, throughout the 32 week program

SECONDARY OUTCOMES:
Health risk assessment | Health risk assessments conducted at baseline, 8 weeks, 32 weeks
  The Health risk assessment includes psychosocial, behavioral (self report), and measured anthropometric and clinical indicators of heart health.
Walking group session attendance | Attendance taken at each session (3 times per week) to determine average weekly attendance; over the 32 weeks
  Attendance at walking group sessions (3times per week) over the 32 week intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Schulz, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States